CLINICAL TRIAL: NCT02790775
Title: Evaluation of the Pain and Visual Outcome Associated With Location of Intravitreal Bevacizumab Injection
Brief Title: Pain and Visual Outcome in Intravitreal Bevacizumab Injection
Acronym: pain & visual
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Ophthalmic Research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 94312
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2015-09

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Injection Anti-VEGF in quadrant 1 (Active Comparator): Each participant receive one injection Anti-vascular endothelial growth factor (Anti-VEGF) in one eye in the quadrant 1
  Interventions: Drug: Anti-VEGF in quadrant 1
- Injection Anti-VEGF in quadrant 2 (Active Comparator): Each participant receive one injection Anti-vascular endothelial growth factor (Anti-VEGF) in one eye in the quadrant 2
  Interventions: Drug: Anti-VEGF in quadrant 2
- InjectionAnti-VEGF in quadrant 3 (Active Comparator): Each participant receive one injection Anti-vascular endothelial growth factor (Anti-VEGF) in one eye in the quadrant 3
  Interventions: Drug: Anti-VEGF in quadrant 3
- InjectionAnti-VEGF in quadrant 4 (Active Comparator): Each participant receive one injection Anti-vascular endothelial growth factor (Anti-VEGF) in one eye in the quadrant 4
  Interventions: Drug: Anti-VEGF in quadrant 4

INTERVENTIONS:
Drug: Anti-VEGF in quadrant 1
  Arms: Injection Anti-VEGF in quadrant 1
Drug: Anti-VEGF in quadrant 2
  Arms: Injection Anti-VEGF in quadrant 2
Drug: Anti-VEGF in quadrant 3
  Arms: InjectionAnti-VEGF in quadrant 3
Drug: Anti-VEGF in quadrant 4
  Arms: InjectionAnti-VEGF in quadrant 4

SUMMARY:
In this double blind clinical trial, 1000 patients suffering from diabetic macular edema, age-related macular degeneration, neovascularization due to proliferative diabetic retinopathy and cystoid macular edema secondary to retinal vascular occlusions are included. Those with the history of Ocular pain prior to the procedure, any contraindication for Intravitreal Bevacizumab Injection (IVI), history of any kind of anterior segment conditions that could affect pain sensation, history of using systemic analgesic or sedative medications, history of previous eye surgery other than for cataract, glaucoma, uveitis and bullous keratopathy and poor cooperation in using the visual analogue scale (VAS) are excluded from the study. Before starting the treatment all patients undergo complete ophthalmic exam , best-corrected visual acuity (BCVA) checking and macular thickness measurements using optical coherence tomography (OCT). Patients are randomly assigned to each group .Each participant receive one injection in one eye in this study. Pain is measured by subjective grading on a Visual Analog Scale (VAS) immediately after IVI. BCVA and OCT would be checked again at month one.

ELIGIBILITY:
Inclusion Criteria:

* diabetic macular edema, age-related macular degeneration, neovascularization due to proliferative diabetic retinopathy and cystoid macular edema secondary to retinal vascular occlusions

Exclusion Criteria:

* history of Ocular pain prior to the procedure, any contraindication for Intravitreal Bevacizumab Injection (IVI), history of any kind of anterior segment conditions that could affect pain sensation, history of using systemic analgesic or sedative medications, history of previous eye surgery other than for cataract, glaucoma, uveitis and bullous keratopathy and poor cooperation in using the visual analogue scale (VAS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05-30 (Actual); Study Completion 2016-08-30

PRIMARY OUTCOMES:
Pain | immediately after Intravitreal Bevacizumab Injection
  Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) | preoperative and 1 month postoperatively.
  using Snellen chart

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Republic of Iran, Tehran, Iran